CLINICAL TRIAL: NCT03003702
Title: Domiciliary Monitoring to Predict Exacerbations of COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16/LO/1120
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: COPD Exacerbation

ARMS (2):
- ETH (Experimental): Overnight monitoring
  Interventions: Device: Nonin
- CTH (Other): Morning monitoring
  Interventions: Device: Nonin

INTERVENTIONS:
Device: Nonin

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a common, long term condition of the lungs that is usually caused by cigarette smoking. In addition to daily symptoms and limitation in activities, patients are prone to developing chest infections called 'exacerbations'. Exacerbations are a big problem: unpleasant for patients, and sometimes severe enough to cause hospital admission (and therefore health facilities pressures) and death. Reducing the impact of exacerbations is very important. Investigators have previously shown that earlier treatment of COPD exacerbations results in faster recovery, and reduced chance of hospital admission. Helping patients to detect exacerbations early is therefore important. Investigators have also recently shown that monitoring heart rate and oxygen saturation via a finger probe may assist in this. However, measuring these variables when the patient is awake means they can be affected by other things, such as exercise and anxiety. Our new idea is that measuring heart rate and oxygen level overnight, when a patient is asleep, will give the best chance of detecting COPD exacerbations early and our study will test that. Investigators will randomly allocate 77 patients with COPD recruited from our service in London to standard monitoring, or overnight monitoring, for up to six months or the first exacerbation, whichever is sooner. Investigators will then analyse whether overnight monitoring was able to detect exacerbations earlier, and therefore could be used to help patients get treatment earlier. A subset of participants will also wear an activity monitor overnight for the first two weeks, so that Investigators can assess the effect (if any) of overnight awake periods (such as trips to the bathroom) on the heart rate and saturation recording.

ELIGIBILITY:
Inclusion Criteria:

1. Patient diagnosed with COPD (smoking history of ≥10 pack years and FEV1/VC < 0.7 post-bronchodilator).
2. Patient who had two or more self-reported moderate or severe COPD exacerbations in the past 12 months.
3. Patient who can use study equipment and attend appointments.
4. Can communicate in English.

Exclusion Criteria:

1. Patient who was diagnosed with obstructive sleep apnea (through a self-report and/or a result of Stop Bang and Epworth questionnaires).
2. Patient with co-morbidity preventing taking part.
3. Patients already involved in an ongoing research study.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the difference in time to receive treatment from exacerbation onset as defined by symptoms, compared to exacerbation onset as defined by change in physiology | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Free Hospital NHS, London, United Kingdom

REFERENCES:
- [Derived] Al Rajeh AM, Aldabayan YS, Aldhahir A, Pickett E, Quaderi S, Alqahtani JS, Mandal S, Lipman MC, Hurst JR. Once Daily Versus Overnight and Symptom Versus Physiological Monitoring to Detect Exacerbations of Chronic Obstructive Pulmonary Disease: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Nov 13;8(11):e17597. doi: 10.2196/17597. PMID 33185560